CLINICAL TRIAL: NCT06808165
Title: Evaluation of Relaxin and Placental Volume in Placenta Accreta Spectrum Disorders: A Case-Control Study
Brief Title: Relaxin and Placental Volume in Placenta Accreta Spectrum
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: KAEK/2023.01.20
Record Dates: First submitted 2025-01-29; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Placenta Accreta Spectrum; Placenta Accreta / Percreta
Keywords: Biomarker; PAS; Placenta Accreta Spectrum; Placental Volume; Relaxin; RLN2
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Human relaxin-2 (RLN2) levels were measured in maternal serum samples stored at 2-8°C before being discarded, using a Human RLN2 ELISA Kit (Sunred Biological Technology, Shanghai, China) as per the manufacturer's instructions before routinely storing maternal venous blood and umbilical cord arterial blood samples were discarded for legal periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Placenta Accreta Spectrum Group: * 20 patients diagnosed with PAS, confirmed through histopathological findings post-cesarean hysterectomy
  * Blood and placental tissue analyzed for relaxin levels and placental volume
  * Subgroup analysis based on PAS severity (accreta, increta, percreta)
  Interventions: Diagnostic Test: relaxin
- Control Group (No PAS Pathology with Elective Cesarean Section): * 20 healthy pregnant women undergoing elective cesarean section
  * Blood and placental volume assessed
  Interventions: Diagnostic Test: relaxin

INTERVENTIONS:
Diagnostic Test: relaxin — The primary source of relaxin in pregnancy is the corpus luteum, but it is also produced in other tissues, such as the decidua and placenta. Importantly, relaxin's pleiotropic effects include endothelial-dependent vasodilation, extracellular matrix remodeling, and potential contributions to placental development. These properties make relaxin a molecule of interest in the context of PAS disorders, where abnormal placental invasion may reflect disruptions in vascular and extracellular matrix regulation. Additionally, recent findings have indicated altCirculating relaxin levels were assessed before routinely storing maternal venous blood and umbilical cord arterial blood samples are anelyzed. This study aimed to compare relaxin levels in umbilical cord and peripheral blood and estimated placental volumes (EPV) between PAS cases and controls. Additionally, subgroup analysis was conducted to evaluate relaxin levels and EPV among PAS subtypes (accreta, increta, and percreta).

SUMMARY:
This retrospective case-control study investigated the potential role of circulating relaxin levels and estimated placental volumes (EPV) in the pathogenesis and diagnosis of placenta accreta spectrum (PAS) disorders. It compared these parameters in patients diagnosed with PAS versus healthy controls.

DETAILED DESCRIPTION:
This study aimed to compare relaxin levels in umbilical cord and peripheral blood and estimated placental volumes (EPV) between PAS cases and controls. Additionally, subgroup analysis was conducted to evaluate relaxin levels and EPV among PAS subtypes (accreta, increta, and percreta).A retrospective case-control study was conducted at a tertiary referral center, analyzing data from January 2022 to December 2022.

ELIGIBILITY:
Inclusion Criteria:

Women aged 18-45 years Confirmed histopathological diagnosis of PAS (case group) Complete medical records Healthy pregnant women undergoing cesarean delivery (control group)

Exclusion Criteria:

Multifetal gestation Emergency surgeries Incomplete medical records

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — * Women aged 18-45 years
  * Confirmed histopathological diagnosis of PAS (case group)
  * Complete medical records
  * Healthy pregnant women undergoing cesarean delivery (control group)
Study Population: The study population consisted of two groups. Following retrospective investigation of patients operated in our clinic between 01.01.2022 and 01.12.2022, the case group included 20 patients diagnosed with PAS disorders, suspected with clinical and imaging findings, confirmed through histopathological findings. These patients had undergone elective cesarean hysterectomy and met inclusion criteria aged between 18 and 45 years and availability of complete medical records. Due to ethical considerations, 4 patients diagnosed with PAS who underwent emergency surgery because of vaginal bleeding and 14 patients operated with segmentary resections were excluded from the study to compose more homogenous study cohort for the measurement of EPV. The control group consisted of 20 healthy pregnant women who underwent the first planned cesarean section of the day, without any obstetric complications, on the same days when planned PAS cesarean-hysterectomy cases were performed in 2022.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Circulating relaxin (RLN2) levels in peripheral and umbilical cord blood | 11 months
  The primary source of relaxin in pregnancy is the corpus luteum, but it is also produced in other tissues, such as the decidua and placenta. Importantly, relaxin's pleiotropic effects include endothelial-dependent vasodilation, extracellular matrix remodeling, and potential contributions to placental development. These properties make relaxin a molecule of interest in the context of PAS disorders, where abnormal placental invasion may reflect disruptions in vascular and extracellular matrix regulation. Additionally, recent findings have indicated altered expression of relaxin, its receptor RXFP1, and insulin-like peptide 4 (INSL4) in PAS cases, suggesting potential roles in its pathogenesis.

SECONDARY OUTCOMES:
placental volume | 11 months
  Placental volume, assessed through imaging modalities, has been explored as a potential biomarker for abnormal placental development, including PAS. Studies have demonstrated that larger placental volumes may be associated with invasive placentation, suggesting a correlation between placental growth patterns and PAS severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Cam and Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burston HE, Kent OA, Communal L, Udaskin ML, Sun RX, Brown KR, Jung E, Francis KE, La Rose J, Lowitz J, Drapkin R, Mes-Masson AM, Rottapel R. Inhibition of relaxin autocrine signaling confers therapeutic vulnerability in ovarian cancer. J Clin Invest. 2021 Apr 1;131(7):e142677. doi: 10.1172/JCI142677. PMID 33561012
- [Background] Ma P, Hu T, Chen Y. The Association and diagnostic value between Maternal Serum Placental Markers and Placenta Previa. Eur J Obstet Gynecol Reprod Biol X. 2024 Oct 11;24:100346. doi: 10.1016/j.eurox.2024.100346. eCollection 2024 Dec. PMID 39483207
- [Background] Patil NA, Rosengren KJ, Separovic F, Wade JD, Bathgate RAD, Hossain MA. Relaxin family peptides: structure-activity relationship studies. Br J Pharmacol. 2017 May;174(10):950-961. doi: 10.1111/bph.13684. Epub 2017 Jan 19. PMID 27922185
- [Result] Goh W, Yamamoto SY, Thompson KS, Bryant-Greenwood GD. Relaxin, its receptor (RXFP1), and insulin-like peptide 4 expression through gestation and in placenta accreta. Reprod Sci. 2013 Aug;20(8):968-80. doi: 10.1177/1933719112472735. Epub 2013 Jan 9. PMID 23302396